CLINICAL TRIAL: NCT01549119
Title: Multicentre, Randomized, Placebo-controlled, Double-blind, Phase I/IIa Dose-escalation Clinical Study of a Therapeutic Vaccine (VAC-3S) Intended to Confer Protection Against Immunopathological Effects of HIV-1 in Infected Patients
Brief Title: Phase I/IIa Dose-escalation Clinical Study of VAC-3S
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InnaVirVax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVVAC-3S/P1
Record Dates: First submitted 2012-03-02; First posted 2012-03-08 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; HIV; immunotherapy; active immunotherapy; vaccine; virulence; innate immunity; NK cells

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Low dose VAC-3S (Experimental)
  Interventions: Biological: VAC-3S
- Medium dose VAC-3S (Experimental)
  Interventions: Biological: VAC-3S
- High dose VAC-3S (Experimental)
  Interventions: Biological: VAC-3S
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Double-dose VAC-3S (Experimental)
  Interventions: Biological: VAC-3S

INTERVENTIONS:
Biological: VAC-3S — Comparison of different doses of vaccine. Liquid form Volume: 0.5 mL - 2 X 0.5 mL for double-dose arm 3 vaccinations at one month apart
  Arms: Double-dose VAC-3S; High dose VAC-3S; Low dose VAC-3S; Medium dose VAC-3S
Biological: Placebo — Comparison with experimental vaccine
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the safety and immunogenicity of the therapeutic vaccine candidate VAC-3S in HIV-1 infected patients under AntiRetroviral Therapy (ART) with undetectable viral loads.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patient
* Age between 18 and 55 years
* ART (AntiRetroviral Therapy) initiation 1 year ago
* Plasma HIV RNA below 50 copies per ml on three sequential occasions including V-1 in the past 12 months
* CD4 T cell count above or equal to 200 cells per mm3,
* Nadir CD4 T cell count above or equal to 100 cells per mm3,
* Contraception in women with child-bearing potential

Exclusion Criteria:

* Any ART change within a month preceding screening.
* Chronic active liver disease, HIV-Hepatitis Coinfection.
* Immunotherapy in the past year, immunosuppressive treatment within the past month.
* History of auto-immune disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of Study Participants Who Tolerated three vaccinations with VAC-3S at 4-weeks apart Determined by Safety Parameter Changes According to the DAIDS (Division of Acquired Immunodeficiency Syndrome) Adverse Events (AE) Grading Table. | from D0 to week 24
  Safety parameters include adverse events, vital signs, physical examinations, laboratory tests (hematology, blood chemistry, viral load).

SECONDARY OUTCOMES:
Anti-3S antibody titers | from D0 to week 60
Number of Study Participants Who Tolerated three vaccinations with VAC-3S at 4-weeks apart Determined by Safety Parameter Changes According to the DAIDS (Division of Acquired Immunodeficiency Syndrome) Adverse Events (AE) Grading Table. | from week 24 to week 60
  Safety parameters include adverse events, vital signs, physical examinations, laboratory tests (hematology, blood chemistry, viral load).
NKp44L expression on the surface of CD4+ T lymphocytes | from D0 to week 60
Markers of progression to AIDS. Markers include CD4+ cell count, viral load, and phenotypic markers of lymphocyte differentiation and activation. | from D0 to week 60

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Ho Tsong Fang, DVM, PHD, Study Director — InnaVirVax
Locations (2):
- France (2):
  - Hopital Pitie Salpetriere, Paris
  - CIC Cochin Pasteur, Paris

REFERENCES:
- See also: Sponsor's website — http://www.innavirvax.fr